CLINICAL TRIAL: NCT05500950
Title: Application of Color Ultrasound Doppler and CT in the Diagnosis of Lacrimal Sac Space-occupying Lesions
Brief Title: Color Doppler Ultrasound in Lacrimal Sac Space-occupying Lesions
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Associate Chief Physician, Wenzhou Medical University
Other Study IDs: CDU in lacrimal sac
Record Dates: First submitted 2022-07-08; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Dacryocystitis; Chronic; Lacrimal Sac Space-occupying Lesions; Color Doppler Ultrasound; Computed Tomography
Keywords: Color Doppler ultrasound; lacrimal sac space-occupying lesions; nasolacrimal duct obstruction; Computed Tomography
MeSH Terms: conditions — Dacryocystitis; Bronchiolitis Obliterans Syndrome; Lacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with space occupying lesions completed CDU and CT-DCG or CT: Patients who had completed CDU and CT-DCG or CT examination before surgery and were diagnosed with lacrimal sac space occupying lesions during surgery were selected to be included in this study.
  Interventions: Other: CDU and CT-DCG or CT examination

INTERVENTIONS:
Other: CDU and CT-DCG or CT examination — patients with space occupying lesions in the lacrimal sac area completed CDU and CT-DCG or CT examination before surgery

SUMMARY:
Dacryocystitis and nasolacrimal duct obstruction are the main common causes of epiphora. Dacryocystorhinostomy (DCR) is a widely used and effective treatment for dacryocystitis and nasolacrimal duct obstruction. Among these cases, some patients have space-occupying lesions in the lacrimal sac area, such as dacryoliths, mucoceles, granulomas, and even tumors. For patients with lacrimal sac tumors, a more complex treatment plan needs to be adopted, and the severity of the disease and the complexity of treatment should be informed before surgery, since more than 55% of lacrimal sac tumors are malignant.

Therefore, preoperative diagnosis and identification of lacrimal sac space-occupying lesions is important. For lack of imaging examinations, and the symptoms of patients with space-occupying lesions are often similar to those of dacryocystitis and nasolacrimal duct obstruction, which lead to the diagnosis of lacrimal sac space-occupying lesions was not discovered before DCR. CDU has been used for the observation of lacrimal gland tumors. This study has attempted to assess the CDU and CT dacryocystography characteristics of the lacrimal sac space-occupying lesions.

DETAILED DESCRIPTION:
A retrospective analysis was performed on the patients with lacrimal sac space-occupying lesions during endoscopic endonasal dacryocystorhinostomy（EEDCR） surgery in the Eye and Optometry Hospital Affiliated to Wenzhou Medical University from January 2018 to March 2022. Patients who had completed color Doppler ultrasound and CT dacryocystography or CT examination before surgery and were diagnosed with lacrimal sac space-occupying lesions during EEDCR surgery were selected to be included in this study. A total of 33 cases of lacrimal sac space-occupying lesions were found, however, preoperative ultrasound or CT examination was absent in 12 of them. Finally, 21 patients were enrolled in this study. We compared preoperative color Doppler ultrasonography and CT dacryocystography or CT examination in these 21 patients according to pathological diagnosis, and recorded the success rate of DCR and the recurrence rate of lacrimal sac space-occupying lesions at follow-up.

CDU was performed in all patients were examined in the supine position. The skin corresponding to the lacrimal fossa region were coated with disinfectant coupling agent, then the probe was placed over the skin and moved in transverse and cranio-caudal directions. A qualitative assessment of the size of the lacrimal sac, sac content, and surrounding structures was first performed in B-mode. Then, color Doppler ultrasound was used to analyze whether there is blood supply in the lacrimal sac space-occupying lesions. CT-DCG images were acquired after injection of a water-soluble iodinated contrast medium through the lower lacrimal punctum, with the layer thickness from 1mm to 5mm.

The fundamental information of all patients is recorded as follows: age, sex, side of involvement, duration of epiphora and history of lacrimal system intervention. All the space-occupying lesions obtained during surgery were sent for pathological examination. All patients were followed up for more than 1 month.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of lacrimal sac space-occupying lesion. Lacrimal sac surgery must be completed. Must had completed color Doppler ultrasound and CT dacryocystography or CT examination before surgery.

Exclusion Criteria:

Preoperative ultrasound or CT examination not completed.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 21 patients who had completed color Doppler ultrasound and CT dacryocystography or CT examination before surgery and were diagnosed with lacrimal sac space-occupying lesions during EEDCR surgery were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Morphological changes of color Doppler ultrasound in lacrimal sac space-occupying lesions | 2 weeks before surgery
  Conventional ultrasonography and color Doppler ultrasonography images are used to assess the characteristics of lacrimal sac space-occupying lesions. Percentage of patients with clear or unclear borders, even or uneven internal echogenicity, regular or irregular shape, with or without blood flow signals of different kinds of lacrimal sac space-occupying lesions was recorded.

SECONDARY OUTCOMES:
Morphological changes of CT or CT-DCG in lacrimal sac space-occupying lesions | 2 weeks before surgery
  2. CT or CT-DCG images are used to assess the characteristics of lacrimal sac space-occupying lesions. Percentage of patients with Regular or irregular shape of different kinds of lacrimal sac space-occupying lesions were recorded. Percentage of the space-occupying lesions in the lacrimal sac invade the surrounding bone was also analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital and School of Ophthalmology and Optometry,Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Personal participant data can be requested by email from the corresponding author
Supporting Information: CSR